CLINICAL TRIAL: NCT03229109
Title: Spectrophon Dehydration Body Monitor Accuracy Evaluation
Brief Title: Analysis of Sweat Secretion and Body Dehydration Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Collaborators: Ariel University (Other)
Responsible Party: Principal Investigator, Anatoly Kreinin, MD, PHD, Head of Psychiatry Department,, Tirat Carmel Mental Health Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 04/17
Record Dates: First submitted 2017-07-05; First posted 2017-07-25 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Dehydration
Keywords: dehydration; spectrophon; device; perspiration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Age 18-25, males and females, Spectrophon dehydration body monitor was attached to subject's wrist
  Interventions: Device: Spectrophon dehydration body monitor
- Group 2 (Experimental): Age 26-35, males and females, Spectrophon dehydration body monitor was attached to subject's wrist
  Interventions: Device: Spectrophon dehydration body monitor
- Group 3 (Experimental): Age 36-45, males and females, Spectrophon dehydration body monitor was attached to subject's wrist
  Interventions: Device: Spectrophon dehydration body monitor
- Group 4 (Experimental): Age 46-50, males and females, Spectrophon dehydration body monitor was attached to subject's wrist
  Interventions: Device: Spectrophon dehydration body monitor

INTERVENTIONS:
Device: Spectrophon dehydration body monitor — Participants (both males and females) were assigned to physical activity (running), biosensor was attached to subject's wrist

SUMMARY:
Monitoring of a person's physical status is a key point for maintaining of "healthy life". Wearable devices provide a unique possibility for real-time monitoring. This study aims to estimate the accuracy of Spectrophon Dehydration Body Monitor (DBM) incorporated in smartwatch Samsung Gear S2 and sport band Samsung Gear Fit2 by comparing data obtained by DBM with the total weight lost during exertion.

DETAILED DESCRIPTION:
Reduced physical activity is considered as a risk factor for obesity, diabetes, cancer and depression. A proper exercise program can mitigate cognitive and physical decline associated with ageing. Existing general guidelines for physical activity are not universal or appropriate for every person. A personalized approach based on a subject age and unique combination of different physiological parameters would serve as a solution for finding optimal training protocols for individuals. Hence, monitoring basic physiological and biochemical parameters and obtaining information reflecting the body metabolic state is necessary for health status estimation to develop the abovementioned personally-oriented training protocols. Dehydration Body Monitor (DBM) developed by Spectrophon L.T.D. can measure sweat lost, salt concentration in sweat, and sweating dynamics, which can be used for personal physical status monitoring. This is important not only for controlling appropriate body hydration level but also for keeping kidneys "healthy". Currently, only few DBM tools are available on the market, so there is a growing need for new effective accurate real-time DBM sensors.

The main objective of current study is to estimate the accuracy of Spectrophon DBM incorporated in smartwatch Samsung Gear S2 and sport band Samsung Gear Fit2. The secondary aim of the study is to evaluate the safety-in-use of Spectrophon DBM.

Tested device:

Name: Dehydration Body Monitor; Source: Spectrophon, L.T.D.; Model: SP-DBM Firmware version: 1.5

4. Experimental Design Healthy adults (n=200) in different age and gender groups were recruited for the study. Samsung Gear S2 smartwatch with Spectrophon DBM attached to the bottom of the smartwatch were placed on the right wrist of each participant. At the same time, Samsung Gear Fit2 sport band with Spectrophon DBM attached to the bottom of the band was placed on the left wrist of the participant. Each participant was subjected to moderate physical activity. Data from Samsung Gear S2 and Samsung Gear Fit2 was obtained simultaneously. In parallel, subject weight was also monitored using commercially available digital balancers (Shekel B-200-P).

The evaluation of the measurement accuracy of the Spectrophon DBM was defined as the difference between subject weight change during the exertion (due to sweating and water consumption) and the volume of sweat detected by Spectrophon DBM.

5. Procedures: Participants were weighed prior to the experiment (no clothing after maximal drying) and then subjected to physical activity (walking on the treadmill).

Total duration of study: 90 minutes

5.2 Intensity of exercises:

Participants could choose high or low intensity of exertion:

1. High: up to 6.5km/h;
2. Low: yo to 6.0km/h; 5.3 Data recording: After DBM application was activated, DBM started recording data (sweat rate and total salt in sweat) every 20 sec. and automatically saved results into archive on a mobile phone linked to Samsung Gear S2 or Samsung Gear Fit2 by Bluetooth. Manual recording of data was conducted during breaks Participants were also weighed during each break (no clothing after maximal drying).

5.4. Drinking During the procedure, subjects could drink up to 500 ml of water. The weight of the bottle was measured and recorded after drinking during breaks. The difference was subtracted to the weight loss calculation.

5.5 Restrictions:

In this experiment, the following was avoided:

1. Urination during test (empty before T0)
2. Weight loss should not exceed 2%

Participants could cancel the experiment at any point of the procedure if desired.

ELIGIBILITY:
Inclusion Criteria:

1. Age: older than 18, both gender.
2. Ability and willingness to sign an informed consent form for participation in the study.

Exclusion Criteria:

1. Presence of cardiologic or vascular disease.
2. Evidence of any other serious medical disorder.
3. Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kreinin, MD, PHD, Principal Investigator — Bruce Rappaport Medical Faculty, Technion, Haifa, Israel
Locations (2):
- Israel (2):
  - Mental Health Center, Tirat Carmel, Haifa District
  - Tirat Carmel Mental Health Center, Tirat Carmel, Haifa District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement. Diabetes Care. 2010 Dec;33(12):e147-67. doi: 10.2337/dc10-9990. PMID 21115758
- [Background] Craft LL, Perna FM. The Benefits of Exercise for the Clinically Depressed. Prim Care Companion J Clin Psychiatry. 2004;6(3):104-111. doi: 10.4088/pcc.v06n0301. PMID 15361924
- [Background] Sternfeld B, Weltzien E, Quesenberry CP Jr, Castillo AL, Kwan M, Slattery ML, Caan BJ. Physical activity and risk of recurrence and mortality in breast cancer survivors: findings from the LACE study. Cancer Epidemiol Biomarkers Prev. 2009 Jan;18(1):87-95. doi: 10.1158/1055-9965.EPI-08-0595. PMID 19124485
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Anastasio P, Cirillo M, Spitali L, Frangiosa A, Pollastro RM, De Santo NG. Level of hydration and renal function in healthy humans. Kidney Int. 2001 Aug;60(2):748-56. doi: 10.1046/j.1523-1755.2001.060002748.x. PMID 11473658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 50 | 50 | 50 | 51
Completed | 50 | 50 | 50 | 50
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Not relevant
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 50 | 50 | 50 | 51 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 50 | 51 | 201
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 26 | 101
  Male | 25 | 25 | 25 | 25 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Israel | 50 | 50 | 50 | 51 | 201

OUTCOME MEASURES:

1. Primary Outcome: Number of Measurements Grouped by Level or Error
Description: Number of measurements obtained with Dehydration Monitor with errors greater/less than 20% (as compared to Shekel B-200-P)
Time Frame: 90 minutes
Measure: Number; unit: Number of measurements
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 50 | 50 | 50 | 50
Number of measurements
  Samsung Gear S2 : <20% errors in measurements | 48 | 48 | 49 | 50
  Samsung Gear S2 : >20% errors in measurements | 2 | 2 | 1 | 0
  Samsung Gear Fit2 : <20% errors in measurements | 47 | 48 | 46 | 49
  Samsung Gear Fit2 : >20% errors in measurements | 3 | 2 | 4 | 1

ADVERSE EVENTS:
Time Frame: 90 minutes
Description: The trial did not involve any invasive treatments or administration of any medications so no serious adverse events were monitored, which explains why the number of participants at risk for Serious Adverse Events and for All-Cause Mortality is zero.
  However, we asked participants to report any discomfort (e.g. allergic reactions) at the place where Samsung watch or band with DBM were worn.
Groups:
- Age 18-25; Age 26-35; Age 36-45; Age 46-50: Spectrophon dehydration body monitor was attached to subject's wrist
Arm/Group | Age 18-25 | Age 26-35 | Age 36-45 | Age 46-50
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03229109/Prot_SAP_000.pdf